CLINICAL TRIAL: NCT01953380
Title: Intervention Study to Evaluate the Importance of Information Given to Patients With Contact Allergy
Acronym: ISICA-13
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Andreas Sonesson, MD PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ISICA-13
Record Dates: First submitted 2013-09-20; First posted 2013-10-01 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Dermatitis, Allergic Contact
Keywords: Intervention Studies; Eczema; Randomized Controlled Trial; Knowledge; Quality of Life
MeSH Terms: conditions — Dermatitis, Allergic Contact; Eczema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- extended information (Active Comparator): Extended information on specific allergy
  Interventions: Behavioral: extended information
- Information according to clin. routine (No Intervention): Information according to clinical routine

INTERVENTIONS:
Behavioral: extended information
  Arms: extended information

SUMMARY:
The purpose of this study is to determine whether extended information given to patients with contact allergy improves knowledge, treatment efficacy and daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected contact allergy
* Age above 18 years
* Participants have given informed consent

Exclusion Criteria:

* Mental or language disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
knowledge | one year after inclusion
  knowledge about specific contact allergies and exposure, assessed by questionnaire, a modified version of Nordic Occupational Skin Questionnaire NOSQ-2002/Long, and patient records.

SECONDARY OUTCOMES:
clinical improvement | one year after inclusion
  assessed by questionnaire, a modified version of Nordic Occupational Skin Questionnaire NOSQ-2002/Long, and patient records.
quality of life | one year after inclusion
  assessed by questionnaire, Dermatology Life Quality Index (DLQI).
effect on daily functioning | one year after inclusion
  assessed by questionnaire, a modified version of Nordic Occupational Skin Questionnaire NOSQ-2002/Long, and Dermatology Life Quality Index (DLQI).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Sonesson, MD PhD, Principal Investigator — Region Skåne, Hudkliniken SUS
Locations (1):
- Hudmottagningen SUS, Lund, Skåne County, Sweden

REFERENCES:
- [Derived] Mossing K, Dizdarevic A, Svensson A, Sonesson A. Impact on quality of life of an intervention providing additional information to patients with allergic contact dermatitis; a randomized clinical trial. J Eur Acad Dermatol Venereol. 2022 Nov;36(11):2166-2171. doi: 10.1111/jdv.18412. Epub 2022 Jul 18. PMID 35794786